CLINICAL TRIAL: NCT00224432
Title: Double-Blind, Parallel, Randomised Study to Investigate the Clinical and Immunological Effects of Oral Administration of Probiotic Bacteria in Infants With Atopic Dermatitis With and Without Cow's Milk Allergy.
Brief Title: Double-Blind, Parallel, Randomised Study to Investigate the Effect of Oral Probiotics in Infants With Atopic Dermatitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Groningen Research Institute for Asthma and COPD (Other)
Collaborators: Numico Research Wageningen, the Netherlands (Unknown)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: METc/99/07/116
Record Dates: First submitted 2005-09-13; First posted 2005-09-23 (Estimated); Last update posted 2006-09-27 (Estimated); Status verified 2006-09

CONDITIONS: Atopic Dermatitis; Atopic Eczema; Infantile Eczema
Keywords: Atopic Dermatitis; SCORAD; probiotics; cytokines; Infant
MeSH Terms: conditions — Dermatitis, Atopic

INTERVENTIONS:
Drug: probiotics: Lactobacillus GG, lactobacillus Rhamnosus

SUMMARY:
To study the effect of supplementation of a hydrolyzed formula with probiotic bacteria on clinical and immunological parameters in infants with AD with and without CMA and to compare effectiveness of different strains of probiotics.

DETAILED DESCRIPTION:
* To determine the effect of supplementation of a hydrolyzed formula with probiotic bacteria on clinical and immunological parameters in infants with AD with and without CMA
* To determine the effect of supplementation of a hydrolyzed formula with probiotic bacteria on clinical and immunological reactivity to cow' milk challenge in infants with AD with CMA
* To compare the effectiveness of different strains of probiotic bacteria in improving clinical and immunological outcome in these infants

ELIGIBILITY:
Inclusion Criteria:

* Term infants fulfilling the Hanifin (1989) criteria for atopic dermatitis

  * Suggestive of CMA (one additional symptom)
  * Scorad index (total) >20 at study entry
  * Below 5 months of age
  * Formula, not breast fed
  * Written informed consent from the parents

Exclusion Criteria:

* • Previous or current use of anti-histamines, oral corticosteroids, probiotics

  * Use of systemic antibiotic or anti-mycotic drugs in the previous 4 weeks
  * Congenital intestinal abnormality (eg. Hirschsprung's disease, intestinal atresia)
  * Other GI disease with intestinal inflammation and/or increased intestinal permeability
  * Skin disorder, not atopic dermatitis
  * Participation in another clinical study

Ages: 0 Years to 5 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 45
Dates: Start 2001-03; Study Completion 2002-09

PRIMARY OUTCOMES:
Significant decrease of SCORAD score in treated infants compared to placebo

SECONDARY OUTCOMES:
IL-4, IL-5 and IFN-gamma production of stimulated peripheral blood mononuclear cells
change in fecal TNF-α and α-1-antitrypsin, urinary EDN
effect on faecal bacteria after probiotics

CONTACTS AND LOCATIONS:
Overall Officials: Eric J Duiverman, MD, PhD, Principal Investigator — Dept of Pediatric Pulmonology, University Medical Center Groningen, The Netherlands; Marianne L Brouwer, MD, Principal Investigator — Dept of Pediatric Pulmonology, University Medical Center Groningen, The Netherlands
Locations (1):
- Beatrix Children's Hospital, University Medical Center Groningen, Groningen, Netherlands

REFERENCES:
- [Result] Brouwer ML, Wolt-Plompen SA, Dubois AE, van der Heide S, Jansen DF, Hoijer MA, Kauffman HF, Duiverman EJ. No effects of probiotics on atopic dermatitis in infancy: a randomized placebo-controlled trial. Clin Exp Allergy. 2006 Jul;36(7):899-906. doi: 10.1111/j.1365-2222.2006.02513.x. PMID 16839405